CLINICAL TRIAL: NCT00005528
Title: Genetics of CVD Risk Factors in Samoans
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5060; R01HL052611 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity; Atherosclerosis

SUMMARY:
To evaluate the role of known genes involved in lipid metabolism on serum lipid and apolipoprotein levels in Samoans residing in American and Western Samoa, who were exposed to the biobehavioral changes of modernization.

DETAILED DESCRIPTION:
BACKGROUND:

Modernizing Samoans are characterized by high levels of certain cardiovascular disease (CVD) risk factors such as extreme adiposity and high prevalences of obesity and hypertension. However, lipid levels in Samoans such as total cholesterol and high density lipoprotein (HDL) cholesterol are not consistent with their obesity and not always consistent with ecological measures of modernization.

DESIGN NARRATIVE:

The cross-sectional study used serum lipid and lipoprotein and dietary data collected in 1994 and 1995 in American and Western Samoa to compare the American and Western Samoans. Quantitative determinations were made of lipid and apolipoprotein levels differences between the two groups. Estimates were made of the effects of dietary intake, body size, and smoking on lipid and apolipoproteins. Cross-sectional analyses were performed on genetic factors influencing lipid and lipoprotein levels. Statistical analyses were conducted to test hypotheses about gene-environment interactions and gene-gene interactions in polynesians from American Samoa and Western Samoa.

Diet, physical activity and body size vary with exposure to the influences of economic modernization and the adoption of non-traditional behaviors. Although adiposity and its central distribution, insulin, blood pressure and dietary cholesterol increase from Western Samoa to American Samoa, saturated fat intakes due to coconuts and cigarette smoking are greater in Western Samoa. Thus, modernization does not produce simple unilineal changes in risk factors. The investigators examined very specific hypotheses, based on the cross-sectional data collected in 1994 and 1995, about the influence of genes on lipids, about genetic interactions on lipids and about concrete environmental and specific gene interactions on lipid outcomes.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-04; Study Completion 2000-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Kamboh — University of Pittsburgh

REFERENCES:
- [Background] Kamboh MI, McGarvey ST, Aston CE, Ferrell RE, Bausserman L. Plasma lipoprotein(a) distribution and its correlates among Samoans. Hum Biol. 2000 Apr;72(2):321-36. PMID 10803663
- [Background] Newman JD, McGarvey ST, Steele MS. Longitudinal association of cardiovascular reactivity and blood pressure in Samoan adolescents. Psychosom Med. 1999 Mar-Apr;61(2):243-9. doi: 10.1097/00006842-199903000-00017. PMID 10204978
- [Background] Galanis DJ, McGarvey ST, Quested C, Sio B, Afele-Fa'amuli SA. Dietary intake of modernizing Samoans: implications for risk of cardiovascular disease. J Am Diet Assoc. 1999 Feb;99(2):184-90. doi: 10.1016/s0002-8223(99)00044-9. PMID 9972185
- [Background] Steele MS, McGarvey ST. Anger expression, age, and blood pressure in modernizing Samoan adults. Psychosom Med. 1997 Nov-Dec;59(6):632-7. doi: 10.1097/00006842-199711000-00013. PMID 9407584
- [Background] Steele MS, McGarvey ST. Expression of anger by Samoan adults. Psychol Rep. 1996 Dec;79(3 Pt 2):1339-48. doi: 10.2466/pr0.1996.79.3f.1339. PMID 9009791
- [Background] DePrince K, McGarvey ST, McAllister AE, Bausserman L, Aston CE, Ferrell RE, Kamboh MI. Genetic effect of two APOA repeat polymorphisms (kringle 4 and pentanucleotide repeats) on plasma Lp(a) levels in American Samoans. Hum Biol. 2001 Feb;73(1):91-104. doi: 10.1353/hub.2001.0006. PMID 11332648
- [Background] Moffett S, Martinson J, Shriver MD, Deka R, McGarvey ST, Barrantes R, Ferrell RE. Genetic diversity and evolution of the human leptin locus tetranucleotide repeat. Hum Genet. 2002 May;110(5):412-7. doi: 10.1007/s00439-002-0715-5. Epub 2002 Apr 4. PMID 12073010
- [Background] McGarvey ST, Forrest W, Weeks DE, Sun G, Smelser D, Tufa J, Viali S, Deka R. Human leptin locus (LEP) alleles and BMI in Samoans. Int J Obes Relat Metab Disord. 2002 Jun;26(6):783-8. doi: 10.1038/sj.ijo.0801996. PMID 12037648
- [Background] Tsai HJ, Sun G, Weeks DE, Kaushal R, Wolujewicz M, McGarvey ST, Tufa J, Viali S, Deka R. Type 2 diabetes and three calpain-10 gene polymorphisms in Samoans: no evidence of association. Am J Hum Genet. 2001 Dec;69(6):1236-44. doi: 10.1086/324646. Epub 2001 Nov 5. PMID 11704924
- [Background] Choh AC, Gage TB, McGarvey ST, Comuzzie AG. Genetic and environmental correlations between various anthropometric and blood pressure traits among adult Samoans. Am J Phys Anthropol. 2001 Aug;115(4):304-11. doi: 10.1002/ajpa.1086. PMID 11471128